CLINICAL TRIAL: NCT00642356
Title: An 8-week, Prospective, Randomized, Double-blind, Double-dummy, Active-controlled, Multi-center Comparison Study of the Effects of Carbidopa/Levodopa/Entacapone Versus Immediate Release Carbidopa/Levodopa on Non-motor Symptoms in Patients With Idiopathic Parkinson's Disease and Demonstrating Non-motor Symptoms of Wearing Off
Brief Title: Carbidopa/Levodopa/Entacapone Versus Immediate Release (IR) Carbidopa/Levodopa on Non-motor Symptoms in Patients With Idiopathic Parkinson's Disease and Demonstrating Non-motor Symptoms of Wearing Off
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CELC200AUS14
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Results first posted 2011-01-11 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2011-02

CONDITIONS: Parkinson's Disease
Keywords: Idiopathic Parkinson's disease; carbidopa/levodopa/entacapone; non-motor symptoms; motor-symptoms
MeSH Terms: conditions — Parkinson Disease | interventions — Stalevo; Levodopa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Carbidopa/levodopa/entacapone (Experimental)
  Interventions: Drug: Carbidopa/levodopa/entacapone
- Immediate release carbidopa/levodopa (Active Comparator)
  Interventions: Drug: Immediate release carbidopa/levodopa

INTERVENTIONS:
Drug: Carbidopa/levodopa/entacapone — Carbidopa/levodopa/entacapone 25/100/200 mg tablets plus placebo immediate release carbidopa/levodopa capsules, administered orally for 8 weeks. Total daily dosage and frequency of dosing for each patient was determined by the investigator and stabilized upon entry into the study.
  Other Names: Stalevo®
  Arms: Carbidopa/levodopa/entacapone
Drug: Immediate release carbidopa/levodopa — Immediate release carbidopa/levodopa 25/100 mg capsules plus placebo carbidopa/levodopa/entacapone tablets, administered orally for 8 weeks. The maximum daily dose is 800 mg. Total daily dosage and frequency of dosing for each patient was determined by the investigator.
  Arms: Immediate release carbidopa/levodopa

SUMMARY:
The purpose of this study is to test the effects of carbidopa/levodopa/entacapone compared to the effects of immediate-release carbidopa/levodopa on non-motor symptoms of end-of-dose wearing off in persons who have Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Be aged 30 to 85 years.
* Be male or female - female patients must be either not of childbearing potential (defined as post menopausal for at least one year or surgically incapable of bearing children), or must be practicing contraceptive methods as outlined in the protocol.
* Have a clinical diagnosis of idiopathic Parkinson's Disease, exhibiting at least 2 of 3 symptoms (rigidity, resting tremor, bradykinesia)
* Have non-motor symptoms of end of dose wearing off i.e., the presence of at least one non-motor symptom of Parkinson's Disease which improves with the next immediate release (IR) carbidopa/levodopa dose as determined by the Quantitative Wearing-Off Questionnaire 9 and investigator's assessment. At least one non-motor item has to show a severity of at least 2 points (of a maximum of 4) and show an improvement of at least 1 one hour after immediate release (IR) carbidopa/levodopa administration. Also there should not have been a deterioration of 1 point or more in another non-motor item.(all criteria must be fulfilled)
* Be taking a stable dose of immediate release (IR) carbidopa/levodopa for at least 21 days prior to randomization at an equivalent total daily dose of immediate release (IR) carbidopa/levodopa between 300 to 800 mg. Dosing should be either 3 to 6 times per day.

Exclusion Criteria:

* Have a previous history of being non-responsive to entacapone or tolcapone treatment or having experienced a serious or severe adverse event(s) which resulted in the discontinuation of treatment from the previous use of entacapone or tolcapone; current treatment with entacapone or tolcapone or discontinued treatment with either therapy or discontinued less than 60 days before randomization;
* Have a history, signs, or symptoms suggesting a diagnosis of secondary or atypical parkinsonism;
* Have unstable Parkinson's Disease requiring frequent booster doses;
* Disabling dyskinesias, indicated by a score of greater than 1 on Unified Parkinson Disease Rating Scale question #32, or a score of greater than 1 on Unified Parkinson Disease Rating Scale question #33;
* Have a history or current diagnosis of psychotic features according to the investigator;

Other protocol-defined inclusion/exclusion criteria applied to the study.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- United States (21):
  - Xenoscience, Inc, Phoenix, Arizona
  - South Coast Health Center, Aliso Viejo, California
  - University of California, Irvine, California
  - Coastal Neurological Medical Group, Inc, La Jolla, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Sunrise Clinical Research, Inc, Hollywood, Florida
  - Charlotte Neurological Services, Port Charlotte, Florida
  - Cotton O'Neil Clinic, Topeka, Kansas
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Neurology, Inc, Columbia, Missouri
  - Dr. John's Mercy Medical Center, St Louis, Missouri
  - Creighton U Medical Center, Dept of Neurology, Omaha, Nebraska
  - Parkinson's Disease & Movement Disorders, Commack, New York
  - Central New York Research Corporation, Syracuse, New York
  - Neurological Care of Central NY, Syracuse, New York
  - Duke University, Durham, North Carolina
  - Neurology Associates, Monroeville, Pennsylvania
  - University of Pittsburg, Pittsburgh, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - University of Texas Medical School, Houston, Texas
  - Scott & White Hospital, Temple, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carbidopa/Levodopa/Entacapone | Immediate Release Carbidopa/Levodopa
Started | 7 | 7
Completed | 5 | 4
Not Completed | 2 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 0 | 3
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carbidopa/Levodopa/Entacapone | Immediate Release Carbidopa/Levodopa | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Customized [Number; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >= 65 years | 6 | 7 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on the Non-motor Score of the Quantitative Wearing-Off Questionnaire 9 Item (QWOQ-9)
Description: The QWOQ-9 is a self-rated questionnaire used to assess motor and non-motor symptoms of Parkinson's disease. The 4 non-motor symptoms are each measured on a five item (0-4) Likert scale, reflecting the severity of the item from "not present" to "very severe". The range of possible score values of the non-motor subscale of the QWOQ-9 is 0 to 16. A higher score indicates greater disability. A negative change score indicates improvement.
Time Frame: Baseline to 15 minutes prior to 2nd dose at Week 8
Population: All subjects that were assessed for efficacy
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Carbidopa/Levodopa/Entacapone | Immediate Release Carbidopa/Levodopa
Number analyzed (Participants) | 7 | 5
Units on a scale | -0.9 (0.90) | -0.2 (2.49)

2. Secondary Outcome: Change From Baseline on the Motor Score of the Quantitative Wearing-Off Questionnaire 9 Item (QWOQ-9)
Description: The QWOQ-9 is a self-rated questionnaire used to assess motor and non-motor symptoms of Parkinson's disease. The 5 motor symptoms are each measured on a five item (0-4) Likert scale, reflecting the severity of the item from "not present" to "very severe". The range of possible score values of the motor subscale of the QWOQ-9 is 0 to 20. A higher score indicates greater disability. A negative change score indicates improvement.
Time Frame: Baseline to 15 minutes prior to 2nd dose at Week 8
Population: All subjects that were assessed for efficacy
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Carbidopa/Levodopa/Entacapone | Immediate Release Carbidopa/Levodopa
Number analyzed (Participants) | 6 | 5
Units on a scale | -1.2 (2.23) | 0.0 (2.00)

ADVERSE EVENTS:
Arm/Group | Carbidopa/Levodopa/Entacapone | Immediate Release Carbidopa/Levodopa
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 4/7 | 1/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Carbidopa/Levodopa/Entacapone (N=7) | Immediate Release Carbidopa/Levodopa (N=7)
Nervousness (General disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Urine colour abnormal (Investigations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.